CLINICAL TRIAL: NCT06898632
Title: KidneyCare Cohort Study: Biologic Interrogation of Sarcopenia in Patients With Renal Cell Carcinoma
Brief Title: KidneyCare Cohort Study (KCC-S)
Acronym: KCC-S
Status: Active, not recruiting | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: HCI133144
Record Dates: First submitted 2022-09-08; First posted 2025-03-27 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Kidney Cancer
Keywords: Health Behaviors; Treatment
MeSH Terms: conditions — Kidney Neoplasms; Health Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood: The blood samples will be drawn by a phlebotomist, research nurse, or trained study personnel. A total of 4 tablespoons of blood will be taken during each blood draw.
  Urine: Participants will take a cup into the restroom and fill it about ¾ full with urine.
  Stool: Participants will be provided with a stool collection kit, instructions, mailing containers, and a sample form. The stool sample can be collected at home, frozen, and mailed to Huntsman Cancer Institute (HCI) or delivered in person.
  Tissue: Samples of tumor, normal kidney, and fat tissue which surrounds the kidney will be obtained. Fat tissue under the skin, omentum (fat apron that drapes over the abdomen) and muscle tissue from one of the existing incision sites will also be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: * Will provide blood, urine, and stool samples as well as CT-derived body composition and performance status assessments during the baseline and follow-up study visits.
  * Will provide tissue samples (kidney, fat, omentum, muscle) during cancer surgery.
  * Will provide follow-up questionnaires.
- Cohort 2: * Will provide blood, urine, and stool samples as well as CT-derived body composition during the baseline study visit.
  * Will provide tissue samples (kidney, fat, omentum, muscle) during cancer surgery.
  * Will provide CT-derived body composition during follow-up.

SUMMARY:
This research study aims to learn how lifestyle factors (e.g., obesity) impact the risk of developing kidney cancer and impact survival after nephrectomy (removal of a kidney). The study team's long-term goals are to learn: 1) How to improve treatment success in future patients by tailoring therapies to each patient's unique biology; and 2) What future patients can do to improve their health after diagnosis. To this end, the study team will collect samples (such as blood and extra tissue from surgery) from patients and store and test these samples. The study team also asks patients about their health behaviors (e.g., diet and physical activity) and well-being before their diagnosis and afterwards by filling out questionnaires.

DETAILED DESCRIPTION:
If patients decide to participate in this study, they will be asked to complete the following assessments:

Health questionnaires: The study team will ask participants to complete this health questionnaire within two weeks before their surgery. The questionnaire will ask information about medical history and health-related behaviors.

Follow-up questionnaires: After participants undergo surgery, the study team will contact participants periodically to ask questions about any symptoms they may be experiencing, as well as current physical activity, diet, and quality of life (this will take about 60 minutes to complete). The study team will contact participants with additional questionnaires about 3-6 months post-surgery, 12 months, 24 months, and 60 months later to learn how to improve cancer treatment and overall health after diagnosis for kidney cancer patients.

Performance status assessments: Various measurements of performance status such as handgrip strength, time up & go test, 6-min walk test, and 30-second chair stand will be taken prior to surgery and during follow-up visits (3-6 months and 12 months).

Blood samples: A blood sample will be requested at baseline, as well as at standard of care follow-up visits about 3-6 months and 12 months later during standard follow-up appointments. The study team will request blood samples again at approximately 2 years and 5 years post-surgery.

Urine samples: A urine sample will be requested at baseline and again about 12 months later.

Stool Samples: A stool sample will be requested at baseline and again about 12 months later.

Tissue samples: During kidney surgery, surgeons remove the cancerous tissue. A portion of the tissues will be used by doctors to further understand participants' treatment needs. If there is extra tissue available, the study team asks to obtain samples of tumor, normal kidney, and fat tissue which surrounds the kidney and is usually removed with the surgical specimen. Only tissue that the pathologists decide is not needed for your diagnosis will be used by the study. The study team also asks for permission to collect fat tissue under the skin (subcutaneous), omentum (fat apron that drapes over your abdomen) and muscle tissue from one of the existing incision sites.

Medical records: Participants will also be asked to give study staff permission to copy and review medical records about cancer diagnosis, treatment, and future health as it pertains to participants' cancer prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Renal Cell Cancer (RCC) stage I-IV
* Undergoing radical nephrectomy (entire kidney resection) or partial nephrectomy
* Patients with or without prior systemic therapy for renal cell carcinoma and > 1 year from systemic therapy for other non-cutaneous malignancy
* Cytoreductive nephrectomy (nephrectomy in the setting of limited metastatic disease)

Exclusion Criteria:

* Does not consent to tissue collection
* Patients with only an MRI abdomen/pelvis within 4 months of surgery will be excluded
* Known biopsy-proven non-clear cell RCC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to clinic 2B at the Huntsman Cancer Hospital
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2029-01-09 (Estimated); Study Completion 2029-01-09 (Estimated)

PRIMARY OUTCOMES:
Percent of Scheduled Assessments Completed | End of Participation (60-months post-surgery)
  Feasibility of the study will be assessed by calculating a percentage of scheduled body composition, performance status measurements, performance status questionnaires and biospecimen collections completed.

SECONDARY OUTCOMES:
Change in Muscle Mass | Pre-operative baseline, and at 3, 6, 12, 24, and 60 months post-surgery.
  Using CT-derived body composition analysis, we will assess the mean change in skeletal muscle mass from the pre-operative baseline through 60-months post-surgery.
Change in Visceral Fat | Pre-operative baseline, and at 3, 6, 12, 24, and 60 months post-surgery.
  Using CT-derived body composition analysis, we will assess the mean change in visceral fat area from the pre-operative baseline through 60-months post-surgery.
Change in Functional Status | Pre-operative baseline, and at 3, 6, 12, 24, and 60 months post-surgery.
  Functional status will be assessed using mean change in handgrip strength measured by hand-held dynamometer from the pre-operative baseline through 60-months post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Sanchez, MD, Principal Investigator — University of Utah
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States